CLINICAL TRIAL: NCT02600130
Title: A Phase, I Prospective, Randomized, Double-Blinded, Placebo-controlled, Trial to Evaluate the Safety and Potential Efficacy of Lomecel-B Infusion Versus Placebo in Patients With Alzheimer's Disease
Brief Title: Lomecel-B Infusion Versus Placebo in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Longeveron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00-0000-01
Record Dates: First submitted 2015-11-02; First posted 2015-11-09 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Cohort 1 (10 subjects) Target dose 20 million Longeveron Mesenchymal Stem Cells (LMSCs) via peripheral intravenous infusion.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells
- Cohort 2 (Experimental): Cohort 2 (10 subjects) Target dose 100 million Longeveron Mesenchymal Stem Cells (LMSCs)via peripheral intravenous infusion.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells
- Cohort 3 (Placebo Comparator): Cohort 3 (5 subjects) Placebo (Plasmalyte A and 1% human serum albumin (HSA)) via peripheral intravenous infusion.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Longeveron Mesenchymal Stem Cells — via peripheral intravenous infusion
  Arms: Cohort 1; Cohort 2
Biological: Placebo — via peripheral intravenous infusion
  Arms: Cohort 3

SUMMARY:
This is a Phase I, prospective, randomized, placebo-controlled, double-blinded study designed to test the safety and efficacy of LMSCs (Longeveron Mesenchymal Stem Cells) for the treatment of subjects with clinically diagnosed Alzheimer's disease.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled clinical trial designed to evaluate the safety and efficacy of LMSCs (Longeveron Mesenchymal Stem Cells) or placebo in subjects with Alzheimer's Disease. Following a successful Safety Run-In Phase, a total of twenty-five (25) subjects will be randomized to (2:2:1) to receive low-dose LMSCs, high-dose LMSCs or placebo. After randomization, baseline imaging, and study product infusion, subjects will be followed up at 2,4,13, 26, 39 and 52 week post study product infusion. Intention-to-treat study population will be used for the purpose of the endpoint analysis and safety evaluations.

ELIGIBILITY:
Inclusion Criteria: All subjects enrolled in this trial must:

* provide written informed consent;
* be 50 - 80 years of age at the time of signing the Informed Consent form;
* have a body mass of 45 - 150 kg;
* at the time of enrollment, be diagnosed with AD in accordance with the NINCDS-AA criteria;
* score between 18 and 24 on the Mini Mental State Examination (MMSE);
* has one (or more) identified adult caregiver who is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language at the study site; either lives with the subject or sees the subject for ≥2 hours/day ≥3 days/week; and agrees to accompany the subject to each study visit;
* blood oxygen saturation ≥93% determined via pulse oximetry;
* have a brain MRI consistent with AD;
* have a PET scan using an FDA-approved tracer (e.g., AMYViD, Vizamyl, or Neuraceq), and which indicates the presence of beta-amyloid plaques in the cerebral cortex, within 5 years of enrollment;
* have normal levels of thyroid hormone (free T4) and thyroid-stimulating hormone (TSH);
* have normal levels of B12 and folate;
* have a designated study partner who will accompany the subject to all clinic visits and participate in the subject's clinical assessments; or
* be living in the community, including in an assisted living facility, but excluding long-term care nursing facilities.

Exclusion Criteria: All subjects enrolled in this trial must not:

* be unable to perform any of the assessments required for endpoint analysis;
* show signs of dementia other than AD, such as from AIDS (Acquired Immunodeficiency Syndrome), CJD (Creutzfeldt-Jakob disease), LBD (Lewy Bodies dementia), CVD (Cerebrovascular dementia), PSP (Progressive Supranuclear Palsy), MCI (multiple cerebral infarctions) or NPH (normal pressure hydrocephalus);
* have any other neurodegenerative disease;
* have a history of a seizure disorder;
* have clinically important abnormal screening laboratory values beyond AD;
* have any conditions that would contraindicate an MRI, such as the presence metallic objects in the eyes, skin, or heart;
* have any conditions that would contraindicate a PET scan;
* have > 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis, or evidence of a prior macrohemorrhage as assessed by MRI;
* be currently using corticosteroids or similar powerful steroidal anti-inflammatory medication (e.g., Prednisone) on a regular basis (exceptions allowed include regular use of steroidal nasal sprays, topical steroids, and estrogen-replacement therapy);
* be active listed (or expected to be listed) for transplant of any organ;
* be an organ transplant recipient;
* have a known hypersensitivity to dimethyl sulfoxide (DMSO).
* have a condition that is projected to limited life expectancy to < 1 year.
* have a sitting or resting systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg at Screening;
* have a history of alcohol or drug abuse within the past 5 years.
* have been diagnosed with malignancy within the past 5 years, with the exception of curatively-treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma;
* be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraception (female subjects must undergo a urine pregnancy test at screening and on the infusion day prior to infusion);
* have any serious illness or any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study;
* have any serious illness or any other condition that, in the opinion of the investigator, may compromise the validity of the study (e.g., signs of stroke, traumatic brain injury (TBI), multiple sclerosis (MS), amyotrophic lateral sclerosis (ALS), and Parkinsonism;
* have participated in any investigational therapeutic or device trial within the past 5 years that the investigator feels would influence or affect the outcome of the study;
* be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial;
* be positive for HIV, Syphilis and Hepatitis C; or
* be positive for Hepatitis B. If the subject tests positive for anti-HBc or anti-HBs, subject must be currently receiving treatment for hHepatitis B prior to infusion and remain on treatment throughout the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate the safety of LMSCs administered to subjects with Alzheimer's disease. | 30 days post infusion
  Incidence of any treatment-emergent serious adverse event (TE-SAE), defined as one or more of the following untoward medical occurrences happening within the first 30 days after infusion.
  * Life-threatening event (e.g., stroke or non-fatal pulmonary embolism).
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity.
  * Results in death.
  * Leads to other clinically significant untoward laboratory test result(s) or medical condition(s), determined per Investigator's judgement (e.g., new clinically asymptomatic brain microhemorrhages).

SECONDARY OUTCOMES:
Preliminary efficacy will be determined by examining for changes in AD status and rate decline as assessed by the following. | At Baseline, 2, 4, 13, 26, 39, and 52 weeks
  * Neurological/neurocognitive assessments. ADAS-Cog 11 (Alzheimer's Disease Assessment Scale-cognitive subscale 11) MMSE (Mini Mental State Examination) NPI (Neuropsychiatric Inventory) UPSIT (University of Pennsylvania Smell Identification Test) GDS (Geriatric Depression Scale)
  * Quality of life assessments. ADCS-ADL (Alzheimer's Disease Cooperative Study Activities of Daily Living) QOL-AD (Quality of Life-Alzheimer's Disease)
  * Blood inflammatory and AD biomarkers. IL-1 IL-6 TGF-β1 TNF-α CRP D-Dimer Fibrinogen ApoE
  * Cerebrospinal fluid (CSF) inflammatory biomarkers. IL-1 IL-6 TGF-β1 TNF-α
  * CSF biomarkers of AD. Tau. Phosphorylated tau. Beta-amyloid.
  * Brain volumetry calculated using MRI, including:
  Hippocampal volume. Ventricular volume. Whole-brain volume.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Brain Matters Research, Delray Beach, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Miami Jewish Health, Miami, Florida

IPD SHARING:
Plan to Share IPD: No